CLINICAL TRIAL: NCT04170582
Title: Patient Registry for Patients With Chronic Subdural Hematoma
Acronym: CSDH-R
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-569
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Hematoma; Subdural Hematoma; Chronic
Keywords: Hemorrhage; Subdural; Chronic Subdural Hematoma; Chronic
MeSH Terms: conditions — Hematoma; Hematoma, Subdural; Bronchiolitis Obliterans Syndrome; Hemorrhage; Hematoma, Subdural, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All admitted patients diagnosed with unilateral or bilateral chronic subdural hematoma are included into this registry after consent. Clinical condition, radiological details, therapy (intervention/medication treatment/conservative) and outcome are documented. Patient follow-up is documented over at least 24 month with focus on neurological condition (NIHSS), cognitive impairment (MoCA) and quality of life (SF-12 ver. 2).

DETAILED DESCRIPTION:
Chronic subdural hematoma (cSDH) is a frequent disease in- predominantly - elderly patients often caused by minor trauma to the bridging veins eventually leading to a collection of old blood in the subdural space over time. Besides age of the patients a number of further risk factors are assumed to favor pathogenesis. Depending on size and location of blood collections diverse neurological symptoms can be seen. Therapy approaches are heterogeneous ranging from conservative treatment with or without medication to surgical treatment. There also is lacking knowledge regarding neurocognitive impairment and effects on quality of life in patients under different therapy regimes.

The prospective patient registry will enclose all patients admitted to the investigator's department diagnosed with cSDH either by MRI or CT scan after informed consent. Medical history, regular medication, social status, radiological findings and neurological examination using NIHSS will be performed at time of inclusion, discharge and follow-up. Additionally, neurocognitive testing and documentation of Quality of Life using MOCA Test and SF-12 will be conducted at different timepoints. Moreover a detailed documentation of therapy strategies is implemented in the study protocol.

With this registry the study group expects to obtain significant data leading to a more standardized and optimized therapy regime and furthermore widening understanding on so far rarely known impact of cSDH on neurocognition and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral chronic subdural hematoma
* patient consent

Exclusion Criteria:

* acute subdural hematoma
* no patient consent
* subdural hygroma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic subdural hematomas (cSDH) are a very common pathological entity particularly in the western countries with an aging population. The estimated incidence in older patients is roughly 300/100,000, which is in contrast to the general incidence of less than 20 per 100,000.
  cSDH patients represent a relevant portion of all patients referred to neurosurgical departments.
  The prognosis of cSDH is generally considered to be good even when surgical intervention is required, however cSDH may still result in significant patient mortality and morbidity.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
National Institut of Health Stroke Scale | 24 Month
  Neurological condition as measured by NIHSS: This tool is used to objectively quantify neurological impairment. The score is composed of 11 items each scoring one specific ability with values between 0 and 4 points. A higher score indicates a higher level of impairment. The maximum score is 42, the minimum scor is 0 indicating no neurological impairment.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | 24 month
  Cognitive status as measured by Montreal Cognitive Assessment (MoCA): This score is used to detect cognitive impairment.It was especially validated to detect mild cognitive dysfunction. MoCA scores range form 0 to 30 points, a score above 25 is considered to be normal.
Short Form 12 ver. 2 | 24 month
  Self-perceived quality of life as measured by Short Form 12 (SF-12 ver. 2): This is a shorter version of the short form 36 and is a patient-reported survey of physical and mental well-being. It consists of 12 items representing 4 physical and 4 mental domains which are aggregated into 2 summary measures: Physical Health (PCS) and Mental Health (MCS). Both scales are transformed to have a mean of 50 and a standard deviation of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Kerim Beseoglu, MD, PhD, Principal Investigator — Neurosurgery, Heinrich-Heine-University Düsseldorf, Medical Faculty
Locations (1):
- Department of Neurosurgery, Heinrich-Heine-University Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No